CLINICAL TRIAL: NCT05353296
Title: Dormir Mejor Study: Randomized Controlled Trial of a Culturally Adapted Digital Program of Cognitive-Behavioral Therapy for Insomnia for Spanish Speaking Latina/o Primary Care Patients
Brief Title: Digital Cognitive-Behavioral Therapy for Insomnia in Spanish Speaking Latinas/os (Dormir Mejor Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Carmela Alcantara, Associate Professor, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAS0318; R01HS024274 (AHRQ)
Record Dates: First submitted 2022-04-15; First posted 2022-04-29 (Actual); Results first posted 2025-05-14 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Insomnia
Keywords: Insomnia; Behavioral Sleep Medicine; Digital Health; Hispanic; Latino; Sociocultural
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: This is a parallel-group, single-site, 2-arm Hybrid trial Type-1 effectiveness-implementation study
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to treatment condition
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Culturally adapted digital cognitive behavioral therapy for insomnia (CBT-I) (Somryst) (Experimental): Somryst is an FDA-authorized digital cognitive behavioral therapy for insomnia (CBT-I) program that has been translated and culturally adapted for Spanish speakers. Group will have access to this culturally-adapted Somryst, along with the usual care provided by their primary care provider, and will be provided a sleep hygiene brochure during group assignment.
  Interventions: Behavioral: Digital cognitive behavioral therapy for insomnia (CBT-I) program; Device: Somryst (culturally adapted)
- Minimally Enhanced Usual Care (mEUC) (Active Comparator): Usual care by their primary care provider and a sleep hygiene brochure. Group will continue their typical standard care with their primary care provider, which may include pharmacotherapy. In addition, we will provide a sleep hygiene brochure during group assignment.
  Interventions: Behavioral: Minimally Enhanced Usual Care (mEUC)

INTERVENTIONS:
Behavioral: Digital cognitive behavioral therapy for insomnia (CBT-I) program — A self-guided digital program of CBT-I (Somryst) that has been culturally adapted for Spanish-language speakers. Somryst is an interactive and tailored mobile-based program modeled on the primary tenets of face-to-face CBT-I. Patients will be asked to complete six cores (main intervention content) during the 9-week intervention period. The cores provide key content across six domains including behavioral (sleep restriction, stimulus control), cognitive (cognitive restricting), educational (sleep hygiene), overview, and consolidation/relapse prevention.
  Arms: Culturally adapted digital cognitive behavioral therapy for insomnia (CBT-I) (Somryst)
Behavioral: Minimally Enhanced Usual Care (mEUC) — A minimally enhanced usual care, which will include usual care by patients' Primary Care Provider and a sleep hygiene brochure.
  Arms: Minimally Enhanced Usual Care (mEUC)
Device: Somryst (culturally adapted) — FDA-authorized digital cognitive behavioral therapy for insomnia (CBT-I) trains your brain for better sleep.
  Arms: Culturally adapted digital cognitive behavioral therapy for insomnia (CBT-I) (Somryst)

SUMMARY:
The primary objective of the proposed study is to examine the effectiveness of a culturally adapted digital program of cognitive behavioral therapy for insomnia (CBT-I) compared to minimally enhanced usual care (mEUC) on primary outcomes: reduction in insomnia symptoms at 9 weeks and 6 months post-intervention, using a standard scale among Spanish-Speaking Latina/o adults with chronic insomnia.

DETAILED DESCRIPTION:
Chronic insomnia is associated with significant public health burden and most adults seek care for insomnia in the primary care setting. While Latina/os are at greater risk for insomnia than non-Hispanic Whites, access to the recommended first-line of treatment, cognitive behavioral therapy for insomnia, is limited especially for Spanish-speakers. Recent advances in health information technology such as self-guided digital health treatments represent an innovative and scalable means to address the supply and demand imbalance that perpetuate mental health care disparities, however its implementation in underserved communities remains elusive. The purpose of this study is to compare the effectiveness of a culturally adapted digital version of Cognitive Behavioral Therapy for Insomnia with minimally enhanced usual care on reduction of insomnia symptoms among Spanish-speaking Latina/os adults with chronic insomnia. The study will also examine barriers and facilitators to implementation, and examine cost-effectiveness of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Insomnia Severity Index Score for moderate insomnia symptoms (score>10 on ISS)
* Spanish-speaking or bilingual (English and Spanish) and self-identify as Hispanic or Latina/o
* Report experience of sleep disturbances for at least 3x/week and for at least 3 months

Exclusion Criteria:

* Pregnancy
* Excessive sleepiness (score>=16 on ESS)
* Caregivers of infants (< 3 months) and/or of adults who require care at night
* Participants who are deemed unable to complete the study protocol due to dementia, severe cognitive impairment, severe medical or mental illness, or active substance use disorder
* Untreated moderate to severe obstructive sleep apnea or self-reported narcolepsy
* Unstable depression or insomnia medication regimen
* Patients who have full-time transportation/moving occupations
* Participation in another treatment/intervention study within the time period of initial baseline until the 6-month follow-up assessments
* Participation in regular night shift work, more than 1x/week, or non-standard sleep patterns

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carmela Alcantara, PhD, Principal Investigator — Columbia School of Social Work
Locations (1):
- Columbia School of Social Work, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon request, we plan to make available a de-identified database that includes ISI data, demographics and comorbidity characteristics of patients in our study.
Supporting Information: Study Protocol, SAP
Time Frame: Within 1 year of publication of trial primary outcome results
Access Criteria: De-identified database

RESULTS

PARTICIPANT FLOW:
Groups:
- Culturally Adapted Digital Cognitive Behavioral Therapy for Insomnia (CBT-I) (Somryst): Somryst is an FDA-authorized digital cognitive behavioral therapy for insomnia (CBT-I) program that has been translated and culturally adapted for Spanish speakers. Participants will have access to this culturally-adapted Somryst, along with the usual care provided by their primary care provider, and will be provided a sleep hygiene brochure during group assignment.
- Minimally Enhanced Usual Care (mEUC): Participants will continue their standard care with their primary care provider, which may include pharmacotherapy. In addition, participants will be provided a sleep hygiene brochure during group assignment.
Period: Overall Study
Arm/Group | Culturally Adapted Digital Cognitive Behavioral Therapy for Insomnia (CBT-I) (Somryst) | Minimally Enhanced Usual Care (mEUC)
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Culturally Adapted Digital Cognitive Behavioral Therapy for Insomnia (CBT-I) (Somryst) | Minimally Enhanced Usual Care (mEUC) | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.0 (12.1) | 52.4 (17.2) | 49.2 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Insomnia Severity Index Score (ISI)
Description: ISI is a 7-item self-report scale measuring insomnia symptom severity in the last 2 weeks; summed score ranges 0-28, increasing score associated with increasing severity.
Time Frame: Baseline to post-intervention (9 weeks)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Culturally Adapted Digital Cognitive Behavioral Therapy for Insomnia (CBT-I) (Somryst) | Minimally Enhanced Usual Care (mEUC)
Number analyzed (Participants) | 3 | 4
score on a scale | -6.7 [-15.4 to 2.0] | -3.9 [-12.5 to 4.7]

2. Primary Outcome: Change in Mean Insomnia Severity Index Score (ISI)
Description: as for outcome 1
Time Frame: Baseline to 6 months post intervention
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Culturally Adapted Digital Cognitive Behavioral Therapy for Insomnia (CBT-I) (Somryst) | Minimally Enhanced Usual Care (mEUC)
Number analyzed (Participants) | 3 | 4
score on a scale | -5.7 [-17.1 to 5.8] | -1.6 [-13.0 to 9.9]

3. Secondary Outcome: Change in Mean Quality of Life Score (Short-Form 12 [SF-12], MCS, Mental Component Score)
Description: Short Form (SF)-12 is a 12-item self-report inventory that generically measures quality of life; yields a measure of global health-related wellbeing as 8 domain-specific subscores on a 0-100 scale, increasing score reflects less dysfunction, impairment, or pain. Reporting change in mean mental health component score.
Time Frame: Baseline to post-intervention (9 weeks)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Culturally Adapted Digital Cognitive Behavioral Therapy for Insomnia (CBT-I) (Somryst) | Minimally Enhanced Usual Care (mEUC)
Number analyzed (Participants) | 3 | 4
score on a scale | 10.8 [5.9 to 15.7] | 0.8 [-4.0 to 5.6]

4. Secondary Outcome: Change in Mean Daytime Sleepiness- Epworth Sleepiness Scale (ESS)
Description: ESS is an 8-item brief self-report scale of daytime sleepiness; summed scores range 0-24, where increasing scores constitute greater sleepiness, and a score > 11 represents elevated daytime sleepiness.
Time Frame: Baseline to post-intervention (9 weeks)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Culturally Adapted Digital Cognitive Behavioral Therapy for Insomnia (CBT-I) (Somryst) | Minimally Enhanced Usual Care (mEUC)
Number analyzed (Participants) | 3 | 4
score on a scale | -2.3 [-6.5 to 1.9] | 0.5 [-3.6 to 4.6]

5. Secondary Outcome: Change in Mean Satisfaction With Care Patient Assessment of Chronic Illness Care (PACIC)
Description: PACIC is a 20-item scale containing 5 subscales, adapted for this trial to measure respondents' receipt of services in regards to insomnia in the past 6 months, 5-point scale, range of 20-100 with increasing score reflecting greater satisfaction with care)
Time Frame: Baseline to post-intervention (9 weeks)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Culturally Adapted Digital Cognitive Behavioral Therapy for Insomnia (CBT-I) (Somryst) | Minimally Enhanced Usual Care (mEUC)
Number analyzed (Participants) | 3 | 4
score on a scale | 17.4 [-20.5 to 55.4] | -8.2 [-41.9 to 25.6]

6. Other Pre Specified Outcome: Change in Mean Sleep Quality Pittsburgh Sleep Quality Index (PSQI)
Description: PSQI is an 18-item questionnaire of sleep quality in the past month, summed scores range 0-21, where scores >5 are associated with poor sleep quality and <5 with good sleep quality)
Time Frame: Baseline to post-intervention (9 weeks)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Culturally Adapted Digital Cognitive Behavioral Therapy for Insomnia (CBT-I) (Somryst) | Minimally Enhanced Usual Care (mEUC)
Number analyzed (Participants) | 3 | 4
score on a scale | -1.0 [-2.6 to 0.6] | -0.7 [-2.2 to 0.8]

7. Other Pre Specified Outcome: Change in Mean Self-reported Wake After Sleep Onset
Description: Wake after sleep onset will be recorded in a 14-day sleep diary and refers to the self-reported total number of minutes participants spent awake after they fell asleep. Range: 24 hours Minimum value = 0 minutes (better) Maximum value = 1440 minutes (worse)
Time Frame: Baseline to post-intervention (9 weeks)
Population: This outcome is not able to be analyzed because data not collected.
Arm/Group | Culturally Adapted Digital Cognitive Behavioral Therapy for Insomnia (CBT-I) (Somryst) | Minimally Enhanced Usual Care (mEUC)
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: Change in Mean Actigraphy Assessed Wake After Sleep Onset
Description: Wake after sleep onset will be measured with 14-days of wrist-actigraphy and refers to the total number of minutes participants spent awake after they fell asleep. Range: 24 hours Minimum value = 0 minutes (better) Maximum value = 1440 minutes (worse)
Time Frame: Baseline to post-intervention (9 weeks)
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Culturally Adapted Digital Cognitive Behavioral Therapy for Insomnia (CBT-I) (Somryst) | Minimally Enhanced Usual Care (mEUC)
Number analyzed (Participants) | 3 | 4
minutes | -2.5 [-38.5 to 33.6] | -4.8 [-10.2 to 0.6]

9. Other Pre Specified Outcome: Change in Mean Self-reported Sleep Onset Latency
Description: Sleep onset latency will be recorded in a 14-day sleep diary and refers to the number of minutes that it takes participants to fall asleep. Range: 24 hours Minimum value = 0 minutes (better) Maximum value = 1440 minutes (worse)
Time Frame: Baseline to post-intervention (9 weeks)
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Culturally Adapted Digital Cognitive Behavioral Therapy for Insomnia (CBT-I) (Somryst) | Minimally Enhanced Usual Care (mEUC)
Number analyzed (Participants) | 3 | 4
minutes | -53.3 [-128.6 to 21.9] | -16.9 [-84.7 to 51.0]

ADVERSE EVENTS:
Time Frame: Up to 6 months
Arm/Group | Culturally Adapted Digital Cognitive Behavioral Therapy for Insomnia (CBT-I) (Somryst) | Minimally Enhanced Usual Care (mEUC)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 0/3 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-18): https://cdn.clinicaltrials.gov/large-docs/96/NCT05353296/Prot_SAP_000.pdf